CLINICAL TRIAL: NCT01047085
Title: Does Cholecystectomy Increase the Esophageal Alkaline Reflux? Evaluation by Impedance-pH Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Ahmet Uyanikoglu, Istanbul University, Istanbul Faculty of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Impedance
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2008-03

CONDITIONS: Cholecystolithiasis; Cholecystectomy; Gastroesophageal Reflux
Keywords: cholecystolithiasis; cholecystectomy; gastroesophageal reflux; impedance pH; The relationship between cholecystolithiasis, cholecystectomy and gastroesophageal reflux by impedance pH-method.
MeSH Terms: conditions — Cholecystolithiasis; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Control group: Impedance pH measurements of healthy controls are performed to compare the results with the study group.
  Interventions: Procedure: impedance pH measurement
- Study group (Experimental): Study group: Pre-operative and post-operative impedance pH measurements are performed to patients in which elective cholecystectomy is planned.
  Interventions: Procedure: impedance pH measurement

INTERVENTIONS:
Procedure: impedance pH measurement — Impedance pH measurement: Impedance-pH is a recently developed technique used to monitor all kinds of reflux (gas, liquid, acides and non-acides), reflux level and the clearance period of the esophagus.

SUMMARY:
Publications with different conclusions are available with regard to the correlations between the cholecystolithiasis, cholecystectomy and gastroesophageal reflux disease (GERD). In this study, the controversial relationship between cholecystolithiasis, cholecystectomy and GERD is discussed through the impedance pH method which started to be used in recent years, a method indicating the gas and liquid (acid and non-acid) gastroesophageal reflux (GER) and esophageal clearance time.

DETAILED DESCRIPTION:
Gallstones are observed among 6-20% of the people in the world and 2 folds in women than in men. The symptomatic treatment of the cholecystolithiasis is the cholecystectomy and it is known that every year in United States of America (USA) more than 750.000 cholecystectomy operations are performed. Usually applied to laparoscopic surgery, in experienced hands with great success, but the application is not without problems and can cause the condition called postcholecystectomy syndrome. Postcholecystectomy syndrome is a heterogeneous condition and may occur depending on many causes. One of the suggested reasons is the increasing gastroesophageal reflux diseases (GER). Publications indicating the increase of GER after cholecystectomy are available.

Relationship between the gallbladder stone and the reflux; whether reflux increases after cholecystectomy is a controversial subject. In current studies, the assessments of reflux are performed by different techniques such as interview, endoscopy and 24-hour pH monitoring. These evaluations are often useful in detecting acid reflux. Whereas it is known that after cholecystectomy alkaline bile reflux may be determined in stomach. Therefore, the determination of bile reflux in esophagus after cholecystectomy is also possible. This situation may be important in terms of esophagus adenocarcinoma, because the esophagus adenocarcinoma generally develops in the basis of Barrett's esophagus and alkaline reflux is accepted to contribute to developing Barrett's esophagus (13).

Bile reflux into the stomach is reported in a rate of 30-100% after stomach surgery and 80-90% after gallbladder surgery. Even though bile reflux is observed in such a high percentage, not every kind bile reflux will damage the gastric and esophageal mucosa. Leaking up into the stomach (reflux), the bile and pancreatic secretions presented in the duodenum content mix up with the hydrochloric acid and pepsin presented in stomach, and thereby damage occurs in the gastric and esophageal mucosa. The continuation of this interaction may develop gastritis, esophagitis.

The increase of alkaline reflux and its importance are known in the development of Barrett's esophagus, which is a component of GER spectrum and which can develop into adenocarcinoma. As a result of research performed on people with cholecystectomy, the risk of developing esophageal cancer has been shown to increase moderately. This is probably duo to the reflux of the bile found in the duodenum content through the esophagus. Nowadays only acid reflux can be determined by the widely used 24-hour pH-meter. The bile-sensitive Bilitec is a difficult method to implement and it is not widely used. Impedance-pH is a recently developed technique used to monitor all kinds of reflux (gas, liquid, acides and non-acides), reflux level and the clearance period of the esophagus.

The purpose of this study: To investigate the relationship between GER, cholecystolithiasis and cholecystectomy by using the Impedance-pH method.

ELIGIBILITY:
Inclusion Criteria:

* Participants 20-80 years old, who would undergo cholecystectomy in the General Surgery Clinic due to gallbladder stones, who did not present GER, gastrointestinal system disorders, serious co-morbidities and who agreed to participate in the study were recruited as patients.
* 10 healthy volunteers 20-80 years old, who did not have peptic ulcer, GER, gallbladder stones, cholestatic liver diseases and who agreed to participate in the study were recruited in the control group.

Exclusion Criteria:

* Those who cannot have Impedance-esophageal pHmeter examinations
* Patients with a history of a previous stomach or esophageal surgeries
* Those with malignancies
* Those with severe cardiopulmonary disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)